CLINICAL TRIAL: NCT06588218
Title: Effect of Daily Fresh Watermelon Consumption on Gut and Cardiometabolic Health in Young Adults With Overweight and Obesity
Brief Title: Effect of Watermelon on Gut and Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Ravi Nagpal, PI, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00005203
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Obesity and Overweight; Dysbiosis
Keywords: Gut Microbiome; Dysbiosis; Diet; Overweight; Obesity; Watermelon; Lycopene; Citrulline; Metagenomic; vascular
MeSH Terms: conditions — Obesity; Overweight; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Watermelon Condition (Experimental): This group will maintain a normal diet supplemented with 2.5 cups (~375 grams, 115 kcals, 0.5g fat, 1.5g fiber, 17,225mcg lycopene, 30.75mg vitamin C) of fresh watermelon daily for six weeks
  Interventions: Other: Watermelon
- Control Condition (Active Comparator): This group will maintain a normal diet supplemented with an isocaloric control snack (Belvita breakfast sandwich; 115 kcals, 1.5g fiber, 4.5g fat, 0mg lycopene, 0mg vitamin C) as well as 12 ounces of water
  Interventions: Other: Belvita Breakfast Sandwich + 12 oz Water

INTERVENTIONS:
Other: Watermelon — 2.5 cups of whole fresh watermelon (~375 grams, 115 kcals, 0.5g fat, 1.5g fiber, 17,225mcg lycopene, 30.75mg vitamin C) of fresh watermelon daily for six weeks
  Other Names: Whole Watermelon; Diced Watermelon
  Arms: Watermelon Condition
Other: Belvita Breakfast Sandwich + 12 oz Water — Belvita breakfast sandwich; 115 kcals, 1.5g fiber, 4.5g fat, 0mg lycopene, 0mg vitamin C) as well as 12 ounces of water
  Other Names: Isocaloric Snack; Breakfast Sandwich; Control Snack
  Arms: Control Condition

SUMMARY:
The goal of this clinical trial is to evaluate the effect of daily fresh watermelon consumption for 6-weeks on gut health, including microbiome diversity, gut barrier and immune function in young adults with overweight and obesity. The main questions it aims to answer are:

1. Will consuming fresh watermelon daily for 6-weeks will improve intestinal barrier health and increase microbiome diversity such as an increased population of beneficial 'probiotic' bacteria when compared to control participants consuming a low-fat snack?
2. Will consuming fresh watermelon daily for six-weeks will improve other health measures, including body-composition, blood pressure, blood vessel function, blood lipid profiles, and measures of inflammation, as compared to control participants consuming a low-fat snack for the same time period?

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 30 years old
* Ability to speak and read in English
* Overweight or Obese Class 1 and 2 (BMI ≥ 25 - 39.9 kg/m2)

Exclusion Criteria:

* Intake of antibiotics in the last 3 months
* Intake of pre/pro/postbiotics in the last 3 months
* Current or past (within the last 6 months) user of tobacco, marijuana, or E-cigarette products
* Cardiovascular disease (will not exclude for hypertension), gastrointestinal disease (ulcerative colitis, celiac, Crohn's disease, diverticulosis, peptic ulcers, small intestinal bacterial overgrowth, short bowel syndrome), neurological (multiple sclerosis, meningitis, recent stroke) or endocrine disorders (uncontrolled thyroid disorders, growth hormone disorders, adrenal gland disorders, uncontrolled diabetes - A1C greater than 9%).
* Food allergy to study foods
* Any allergy to melon
* Any allergy to the isocaloric snack (gluten)
* Regular consumption of watermelon greater than 2 servings / week
* Current heavy alcohol use (≥ 15 drinks / week for men, ≥ 8 drinks / week for women
* Class 3 Obesity (BMI > 40 kg/m2)
* Current user of Citrulline, Arginine, Nitric Oxide or other supplements known to affect nitric oxide synthesis (beet root juice or any beet supplement, Pycnogenol / Pine bark extract)
* Known to be currently pregnant (self-disclosed)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Gut Microbiome Diversity | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Collected fecal samples will be used to determine microbiome profiles, including diversity and composition of bacteria.
Change in Oral Microbiome Diversity | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Oral swab samples are collected to determine oral diversity and composition of bacteria in the mouth before and after intervention.

SECONDARY OUTCOMES:
Change in Gut Transit Time | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate changes in gut transit time after watermelon or control snack consumption from baseline to final analysis, using a blue-dye capsule.
Change in Arterial Stiffness | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate the effects of watermelon on arterial stiffness, determined by measuring Pulse Wave Analysis (PWA) and Pulse Wave Velocity (PWV). These are captured by the SphygmoCor XCEL System through the descending aorta to the femoral artery. The aortic pulse wave velocity is detected from carotid and femoral arterial pulses measured non-invasively and simultaneously
Change in Endothelial Function | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate the effects of watermelon on macrovascular endothelial function, which will be evaluated using the flow-mediated dilation (FMD) technique using a Finapres device, which measures the arterial dilation response following acute occlusion of the brachial artery.
Change in Ambulatory Blood Pressure | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate the effect of watermelon on ambulatory blood pressure (systolic and diastolic), determined using a 12-hour ambulatory blood pressure monitor (TM-2440). The 12-hour ambulatory blood pressure monitor will collect blood pressure readings every 20 minutes during waking hours only.
Change in Waist and Hip Circumference | Screening, Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate changes in waist and hip circumference (centimeters), as well as waist-hip ratio at each study visit before, after and during watermelon consumption.
Change in Body Composition | Screening, Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate changes in body composition, including lean mass (kg), fat mass kg), and total body water (kg). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during watermelon consumption.
Change in Habitual Dietary Intake | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Assess changes in habitual dietary intake via 3-day food logs, analyzed using nutrient analysis software.
Change in Biomarkers of Inflammation | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Relevant biomarkers are to be collected via venous blood samples to determine changes in inflammation, including but not limited to C-reactive protein (CRP), IL-1 (Interleukin-1), IL-1 beta, IL-6, IL-10, IL-17, IL-23, Tumor Necrosis Factor Alpha (TNF-a), Interferon-gamma (IFN-Y). All will be expressed in units of pg/mL.
Change in Biomarkers of Appetite | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Relevant biomarkers are to be collected via venous blood samples to determine changes in appetite including Insulin, Glucagon, glucagon-like peptide 1 (GLP-1), Adiponectin, Leptin, Ghrelin, and Peptide YY. All will be expressed in units of pg/mL.
Change in Biomarkers of Intestinal Barrier Function | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Relevant biomarkers are to be collected via venous blood samples to determine changes in intestinal barrier function including LPS (lipopolysaccharides), LBP (lipopolysaccharide binding protein), CD14, Secretory IgA. All will be expressed in units of pg/mL.
Change in Biomarkers of Cardiometabolic Health | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Relevant biomarkers are to be collected via venous blood samples to determine changes in cardiometabolic health including HDL, LDL, total cholesterol, and triglycerides. All will be expressed in units of mg/dL.
Change in Recent Dietary Intake | Screening, Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Assess changes in dietary intake via 24 hr recalls, analyzed using nutrient analysis software.
Change in Body Weight | Screening, Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate changes in body weight (kg) at each study visit before, after and during watermelon consumption.
Change in Body Mass Index | Baseline (day 0), Visit 2 (week 6), Visit 3 (week 10), Visit 4 (week 16).
  Evaluate changes in Body Mass Index (kg/m2) before, during and after consumption of watermelon.

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Nagpal, PhD, Principal Investigator — Florida State University
Locations (1):
- Florida State University - Gut Biome Lab, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified IPD will not be retain past three years, at the time of this submission the researchers does not plan to make IPD available